CLINICAL TRIAL: NCT04708704
Title: Investigation of Photodegraded Edible Food Dyes in Drinking Water on Thyroid Function
Brief Title: Photodegraded Edible Food Dyes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to start the study due to COVID,
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2000026634
Record Dates: First submitted 2020-12-21; First posted 2021-01-14 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Thyroid; Functional Disturbance
MeSH Terms: conditions — Thyroid Diseases | interventions — Erythrosine; Drinking Water; Iodine

STUDY DESIGN:
Intervention Model Description: The effects of three interventions will be investigated:
  1. Erythrosine, prepared in drinking water (0.69 mg/kg bw/day)
  2. SODIS-treated erythrosine, prepared in drinking water (0.69 mg/kg bw/day)
  3. Iodine, prepared in drinking water 0.075 mg/kg bw/day)
  The erythrosine and iodine (control exposure) will be prepared in 500 mL of drinking water and participants will received single daily doses for 14 days. This protocol will be repeated for the three subsequent exposure weeks which will be spaced 2 weeks a part. Instead of receiving daily doses of erythrosine, participants will be given 500 mL of water containing photobleached erythrosine or iodine. The spacing between treatment weeks will serve as a washout period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Erythrosine, prepared in drinking water (Experimental): One point-of-use technology in development that has demonstrated potential for inactivating viruses in drinking water is the application of an edible photosensitizing dye to the water for disinfection. When exposed to sunlight, the photosensitizing dye produces singlet oxygen, a reactive oxygen species capable of inactivating a wide range of viruses. Erythrosine, an FDA-approved dye, has proven its ability to disinfect drinking water, achieving 4-log inactivation of bacteriophage MS2 in under 10 minutes of sunlight exposure. Furthermore, the dye photobleaches upon exposure to light, and the accompanying distinct color change (e.g., red to transparent) occurs at a rate comparable to the disinfection, providing a safety indication that disinfection has completed, a much-needed function lacking in other point-of-use technologies.
  Interventions: Dietary Supplement: Erythrosine, prepared in drinking water (0.69 mg/kg bw/day); Dietary Supplement: SODIS-treated erythrosine, prepared in drinking water (0.69 mg/kg bw/day); Dietary Supplement: Iodine, prepared in drinking water 0.075 mg/kg bw/day)

INTERVENTIONS:
Dietary Supplement: Erythrosine, prepared in drinking water (0.69 mg/kg bw/day) — Erythrosine will be obtained from Roxy & Rich Inc. (Intense Water-Soluble Food Colorant - Pink), which is certified to be edible and complies with US FDA, Health Canada, and European food safety standards. The erythrosine will be prepared in 500 mL of drinking water and participants will received single daily doses for 14 days. We will use a targeted dose of 0.69 mg/kg bw.
Dietary Supplement: SODIS-treated erythrosine, prepared in drinking water (0.69 mg/kg bw/day) — Erythrosine will be SODIS-treated to produce photobleached erythrosine. Transparent 500 mL polyethylene terephthalate (PET) plastic water bottles will be commercially purchased (Kirkland Signature Purified Water). All branding information and labeling will be removed from the bottles. Water bottles will be dosed with ~41 mg erythrosine (0.69 mg/kg bw) using an erythrosine stock solution (8.2 g/L) and will be shaken to mix. The erythrosine-dosed bottles will be placed on a metal shelf and exposed to natural sunlight on the roof of Yale Engineering. Sunlight exposure will be conducted until the absorbance value of erythrosine at the absorption maximum of 526 nm falls below 0.05 above baseline, as measured by ultraviolet-visible spectroscopy. The water bottles containing photobleached erythrosine will be stored under refrigeration in the dark until consumption by participants.
Dietary Supplement: Iodine, prepared in drinking water 0.075 mg/kg bw/day) — Iodine used in the study will be in the form of FCC-grade potassium iodide, which will be obtained from VWR. FCC grade potassium iodide meets the requirements set by the Food Chemical Codex and is suitable for all applications in foods and beverages. Iodine (control exposure) will be prepared in 500 mL of drinking water and participants will received single daily doses for 14 days. We will use a targeted dose of 0.75 mg/kg bw.

SUMMARY:
Assess and contrast the effect of erythrosine and photodegraded erythrosine on thyroid function. Thyroid function will be evaluated as serum triiodothyronine (T3), thyroxine (T4), thyroid stimulating hormone (TSH), T3 resin uptake as well as measures of iodine in serum and plasma before and after a 14-day repeat administration of these edible dyes in drinking water. Dose-related increases in serum and plasma-bound iodine are expected for both erythrosine and photodegraded erythrosine over the 14-day exposure period. TSH is also expected to increase following repeat administration of erythrosine and photodegraded erythrosine. Erythrosine and photodegraded erythrosine are expected to induce an equivalent dose-response increase in thyroid function-related hormone levels.

DETAILED DESCRIPTION:
Access to safe drinking water is a fundamental human right recognized by the United Nations, yet achieving universal access in the developing world has been impeded by insufficient water treatment infrastructure and lack of sustained maintenance. As of 2015, 844 million individuals in low- and lower-middle-income countries (LMICs) did not have access to improved drinking water sources and 159 million people directly used untreated surface water, resulting in the loss of 502 thousand lives annually by diarrheal diseases from pathogen-contaminated water. Because drinking water inequity and the associated mortality disproportionally burden the rural developing world, the provision of improved point-of-use (POU) water treatment technologies that are low cost, simple, and require minimal infrastructure is crucial for achieving ubiquitous access to safe drinking water.

Several POU water treatment methods are currently applied in LMICs (e.g., solar disinfection (SODIS), granular media or ceramic pot filtration, chlorination, etc.). Although effective against bacteria, most perform relatively poorly for virus removal, and all POU technologies demonstrate lower efficacy in the field due to compromised initial water quality and operation by relatively unskilled users. While POU technologies have contributed to the reduction of bacterial and parasitic gastroenteritis, instances of viral gastroenteritis have not declined, with viral agents observed in 43% of developing world diarrheal cases.

One POU technology in development that has demonstrated potential for inactivating viruses in drinking water is the application of an edible photosensitizing dye to the water for disinfection. When exposed to sunlight, the photosensitizing dye produces singlet oxygen, a reactive oxygen species (ROS) capable of inactivating a wide range of viruses. Erythrosine, an FDA-approved dye, has proven its ability to disinfect drinking water, achieving 4-log inactivation of bacteriophage MS2 in under 10 minutes of sunlight exposure. Furthermore, the dye photobleaches upon exposure to light, and the accompanying distinct color change (e.g., from erythrosine red to transparent) occurs at a rate comparable to the disinfection, providing a safety indication that disinfection has completed, a much-needed function lacking in other POU technologies. At a total cost of $0.002-0.003 per liter of treated water, it is cheaper than boiling water in several developing nations and is a financially viable water disinfection technology.

Erythrosine, also known as FD&C Red No. 3 in the USA, is approved by the FDA for use in foods, drugs, and cosmetics, with an acceptable daily intake (ADI) of 2.5 mg/kg bw/day. The concentration recommended by literature for disinfection in drinking water is 5.0 µM erythrosine, or approximately 4.4 mg/L. With the average American consuming 2.38 L of drinking water and beverages per day, a daily exposure of 10.5 mg erythrosine/day is expected. Assuming the total water consumption per day in LMICs matches the American consumption of 2.38 L, then a 60-kg individual would experience a daily erythrosine dose of 0.17 mg/kg bw/day, well below the established FDA ADI.

The motivation for investigating the human health effects of erythrosine stems from the unknown behavior of the photodegradation products. While the molecular structure of erythrosine will change upon oxidation by singlet oxygen, the typical reactions of singlet oxygen are addition reactions that do not typically lead to cleavage of the molecular structure. As a result, it is not expected that the absorption rates of erythrosine to change significantly upon oxidative photobleaching. However, these oxidative products have not been previously tested for toxicity and should be examined before allowing erythrosine-based water disinfection to be further developed. Recent tests have attempted to characterize the photooxidation products of erythrosine but were inconclusive.

Furthermore, previous literature states that ~19% of iodine in the molecular structure of erythrosine is released to the solution after exposure to light and oxidation by singlet oxygen. If the previous water treatment parameters are followed (5.0 µM erythrosine, 2.38 L water/day, 60 kg individual), the daily consumption of iodine released from erythrosine would be 1.1 mg I/day. The lowest observed adverse effect level (LOAEL) and no-observed adverse effect level (NOAEL) for iodine are 1.7 mg I/day and 1.0-1.2 mg I/day, resulting in the tolerable upper intake level (UL) of 1.1 mg I/day. If the literature-reported release of iodine from erythrosine is correct, then exposures are at the UL for iodine. Due to the poor absorption of erythrosine by the gastrointestinal tract, it is not expected that the iodine which remains bound to erythrosine to significantly impact the total iodine consumption. While it is not expected that erythrosine-based water treatment to result in adverse outcomes due to exposure to erythrosine photoproducts or overexposure to iodine, it is important to follow a cautious approach and test for its impact before allowing for the further development of a technology that would be consumed daily by individuals in the developing world.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled at Yale University;
* Be 18 years of age or older;
* Be a non-smoker and not be using any contraindicated drugs; and,
* Have no pre-existing health problems.

Exclusion Criteria:

* Not fluent in English.
* Pregnant
* Diagnosis of a thyroid-related disease.
* Levels of TSH, T3 and T4 outside the normal range.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Thyroid Panel | 15 days
  triiodothyronine (T3), thyroxine (T4), thyroid stimulating hormone (TSH) and T3 resin uptake (T3RU) in serum
Complete blood count (CBC) | 15 days
  Whole blood

SECONDARY OUTCOMES:
Iodine | 15 days
  Serum and urine

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No